CLINICAL TRIAL: NCT06467578
Title: Feasibility and Acceptability of 6-week Repeated Measures of Resting Metabolic Rate Using a Portable Indirect Calorimeter
Brief Title: RMR Monitoring Feasibility and Acceptability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Sarah Purcell, Assistant Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H23-03165
Record Dates: First submitted 2024-05-13; First posted 2024-06-21 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Metabolism; Obesity; Weight Loss
Keywords: resting metabolic rate; portable indirect calorimeter; feasibility; acceptability
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Breezing Portable Indirect Calorimeter (Other): Use Breezing to assess RMR once a week for six weeks
  Interventions: Device: Breezing Portable Indirect Calorimeter

INTERVENTIONS:
Device: Breezing Portable Indirect Calorimeter — Indirect calorimeter with face mask and smartphone compatible application

SUMMARY:
Obesity is a leading risk factor for chronic diseases such as type 2 diabetes, cancer, and cardiovascular disease. Generic weight management programs that target dietary intake and physical activity have been shown to be ineffective in maintaining weight loss beyond a 6-month period. Personalizing weight management programs produces more weight loss than generic programs, possibly through improved self-efficacy (confidence in one's ability to control weight through behavior). One way to personalize diet goals for individuals is by resting metabolic rate (RMR; 'metabolism'). This study will explore adherence and satisfaction of 6-weeks repeated at-home measures of metabolism using a portable device in healthy adults with and without obesity. Relationships among adherence and satisfaction outcomes to health behavior variables will be explored using dietary recalls, exercise monitors and questionnaires. Investigators will conduct a 6-week, one-arm feasibility study in order to address these questions. Twenty men and women ages 19-65 will be recruited (up to n=25 participants), among which 10 participants will have a body mass index (BMI) of ≥30kg/m2 (classified as having obesity), and the remaining 10 participants will have a body mass index (BMI) of < 29.9kg/m2 (classified as not having obesity). The baseline study visit will evaluate participant's anthropometric measures, RMR using the ParvoMedics TrueOne 2400 and Breezing indirect calorimeters, psychological and behavioural related parameters. An activPAL device will be provided to measure participant physical activity. Completion of a 3-day diet record following the baseline study visit, in which participants keep a record of all food and beverages consumed over 2 weekdays and 1 weekend, is required. Participants will be asked to use the Breezing device from home to measure their RMR one time/week on the same day of the week (± one day) and at the same time each morning for six consecutive weeks following the baseline visit. A weekly Qualtrics survey will be sent to participants to monitor adherence. A follow-up visit after the six weeks will assess participant's body composition using a Dual X-ray Absorptiometry (DEXA), in addition to completion of a user satisfaction interview with a study team member for descriptive analysis. The measures taken at the baseline study visit will be repeated at the follow-up visit.

DETAILED DESCRIPTION:
Study visits:

Participants will be asked to refrain from food and calorie- or caffeine-containing beverages for at least 12 hours, alcohol for at least 24 hours, and vigorous-intensity exercise for at least 48 hours before each study visit.

Baseline study visit (~3-3.5 hours):

Prior to the baseline study visit, participants will meet with a member of the study team to review the consent form to establish participation status. Participants will be required to confirm their body weight using a digital scale. Participants will then be randomized using online software (http://www.randomization.com) in a 1:1 fashion for the order of RMR measurement device (i.e., starting with Breezing than Parvo or vice versa). RMR will be measured with the Parvo for 15-20 minutes after a period of 25-30 minutes of quiet rest. RMR will be measured with the Breezing for 6-10 minutes using the Breezing mobile application. In addition, participants will be provided a series of validated and standard questionnaires to assess psychological and behavioural related parameters during this visit. Finally, participants will be asked to create an account for the Breezing mobile application, will be provided with a activPAL activity monitoring device, and will be instructed as to how to complete the 3-day diet record.

Follow-up study visit (~3-3.5 hours, 6-8 weeks post baseline visit):

Repeat measures will be taken for body weight, RMR (using both devices), and behavioural questionnaires. In addition, Dual X-ray absorptiometry (DEXA; Hologic Model A) will measure participant's fat-mass, fat-free mass, body fat percentage and bone mineral density. Body composition variables will be expressed in absolute terms and controlling for height (e.g., FM index: FM [kg]/height [m2]); FFM will also be expressed in relation to FM (FM:FFM). Study team members will then conduct 5-10-minute user satisfaction interviews, where participants will be asked to comment on a few open-ended statements. The interviews will be descriptively examined and will not be analyzed in-depth or used to create themes.

Repeated RMR assessment (~20-30 minutes/week, for six consecutive weeks post baseline study visit):

Participants will be instructed to use Breezing one time/week on the same day of the week (± one day) and at the same time each morning for six consecutive weeks. Participants will be asked to use Breezing after a night of their typical sleep quality and quantity, immediately after waking while lying down and in a fasted state. Participants will send weekly Breezing measurements to study team via email. Breezing RMR results will be recorded in secure OneDrive, separate from personal identifying data and the email and pdf will be deleted. If the participants Breezing RMR values are outside of an error range of 15% lesser or greater than baseline values for two consecutive weeks a study team member will email the participant to check if the RMR measurement protocol is being adhered to and possibly schedule a Zoom call with study team member using UBC secure Zoom link to review the Breezing device measurement protocol. Each week participants will be emailed a link to a Qualtrics survey as a weekly check-in for measurement adherence. On weeks 1, 3 and 6 participants will be asked to complete the Systems Usability Scale 47 to assess the usability of the Breezing device and Breezing mobile application.

Physical activity behaviour:

Physical activity will be quantified using activPAL activity monitors (PALTechnologies: Glasgow, Scotland) worn on the mid-thigh for seven days after the baseline study visit and for seven days before the follow-up study visit. This device is a type of accelerometer that records information about time spent sitting, lying, standing, and stepping. Data on total step count, time spent in activities of different intensities, sedentary time, and sleep time will be delineated using the activPAL software, PALanalysis. Participants will be asked to track time in bed and napping, exercise and activPAL removal (if applicable) to help interpret the data.

Feasibility and acceptability outcomes will be assessed using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-65 years
* Ability to read, understand, and speak in English
* BMI over 18.5
* Live within a 1-hour radius of UBCO
* Sedentary or recreationally active, defined as: <300-minutes per week of self-reported voluntary exercise at moderate intensity or greater over the past 12-weeks
* Not currently pregnant or lactating, not planning to become pregnant in the next 12 weeks
* Ability to attend two in-person sessions at UBCO
* Ability and willingness to fast for 12 hours before each study day visit and at least once a week before completing RMR measures using the portable indirect calorimeter
* Access to a mobile device (i.e., smartphone or tablet) with reliable Bluetooth and Wi-Fi connection for the 6 week study duration
* If applicable:
* For people who occasionally (i.e., <1x/day) use cannabis (including cannabidiol-based products): ability and willingness to abstain from cannabis for two days prior to each study day visit, and the morning of each study visit.
* For people who use cannabis daily: ability and willingness to continue to use the exact same amount of cannabis as they normally use for two days prior to each study day visit, the morning of each study visit (if applicable), and during the 6 week study duration.

Exclusion Criteria:

* Current or previous major comorbidities, by self-report, including:
* Cardiovascular disease
* Diabetes (type 1, type 2, pervious gestational)
* Cancer
* Thyroid diseases
* Human immunodeficiency virus or hepatitis B or C
* Renal diseases
* Polycystic ovary syndrome
* Uncontrolled/untreated, by self-report:
* Hypertension
* Dyslipidemia
* Sleep disorders
* Severe depression
* Any other condition that may affect energy balance
* Currently or in the past six months:
* Use of regular medication that may affect energy balance, or sleep
* Regular use of tobacco or nicotine products
* Starting any new prescription medication within two weeks of the first study day visit or planning to do so during the study
* Working night shifts or traveling across more than two time zones within two weeks of and throughout the study
* History of surgical procedure for weight loss at any time (e.g., gastroplasty, gastric bypass, gastrectomy or partial gastrectomy, adjustable banding, gastric sleeve); history of extensive bowel resection for other reasons
* Current alcohol or substance abuse (score ≥ 15 on the Alcohol Use Disorders Identification Test (AUDIT) 32
* Current or past history of eating disorders including anorexia nervosa, bulimia, binge eating disorder (self-report or score >20 on the Eating Attitudes Test - 26 (EATS-26) questionnaire) 33
* Current symptoms of depression (score ≥ 10 on the Center for Epidemiological Studies Depression Scale, 10-item version (CES-D-10))34
* Weight loss >5kg in past 12 weeks for any reason
* Weight loss of >20 kgs in past 3 years for any reason
* Degree or previous work experience (in the past 10 years) in fields highly related to energy balance (e.g., those exercise or nutrition)

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Adherence | 6 weeks
  Qualtrics survey
RMR (portable indirect calorimeter - BreezingTM) | 6 weeks
  Using Breezing device
Satisfaction & feedback (feasibility) | 6 weeks
  In-person interview

SECONDARY OUTCOMES:
Resting metabolic rate (RMR) - metabolic cart indirect calorimeter | 6-8 weeks
  Using Parvo device
Dietary intake | 3 days
  Record of all food and beverages consumed
Physical activity (accelerometry-derived patterns in moderate-to-vigorous activity) | 7 days post-baseline and 7 days pre-follow-up
  Using activPAL device
Self-regulation | 6-8 weeks
  Exercise and Eating Self-Regulation Questionnaire (Exercise 350-420; Diet 10-50, optimal outcome is subjective)
Eating behaviours | 6-8 weeks
  Three-Factor Eating Questionnaire Revised 18-item version (TFEQ-R18, Cognitive restraint 6-24; Uncontrolled eating 9-36; and Emotional eating 3-12, optimal outcome is subjective)
Subjective physical activity | 6-8 weeks
  Leisure Time Exercise Questionnaire (0-21, Higher scores indicate better outcome), Barriers Self-Efficacy Scale (BARSE, 0-130, higher scores indicate better outcome) (responses to multiple questionnaires will be considered in assessing this outcome)
Weight management knowledge questionnaires- Obesity knowledge | 6-8 weeks
  Obesity Knowledge Questionnaire (percentage correct; 0-100%, higher scores indicate better outcome)
Weight management knowledge questionnaires- Physical activity knowledge | 6-8 weeks
  Physical Activity Knowledge Questionnaire (Level 1 1-5; Level 2 0-12; Level 3 no min max values; Level 4 1-5, optimal outcome is subjective)
Body weight | 6-8 weeks
  Digital scale (Min dependant on hight (Min BMI = 18.6), no Max, optimal outcome is subjective)
Weight management knowledge questionnaires- Nutrition knowledge | 6-8 weeks
  Weight Management Nutrition Knowledge Questionnaire (percentage correct; 0-100%, optimal outcome is subjective)
Weight management knowledge questionnaires- Health beliefs and weight efficacy | 6-8 weeks
  Compensatory Health Beliefs Scale (17-102, optimal outcome is subjective), Weight Efficacy Lifestyle Questionnaire (WELQ, 0-200, higher scores indicate better outcome) (responses to multiple questionnaires will be considered in assessing this outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia - Okanagan Campus, Kelowna, British Columbia, Canada